CLINICAL TRIAL: NCT05974917
Title: Serious gaMe Come Interventi Emergenti di E-health Per i Giovani Con distuRbi neuroLogici o rEspiratori (SMILER) - Progetto@Cnr
Brief Title: Serious gaMes as Emerging E-health Interventions for Young People With neurologicaL or rEspiratory disoRders
Acronym: SMILER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istituto di Farmacologia Traslazionale - sede di Palermo, Consiglio Nazionale delle Ricerche (CNR) (Network)
Responsible Party: Sponsor
Other Study IDs: Verbale N° 01/2023
Record Dates: First submitted 2023-06-06; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Serious Game; Asthma in Children; Children, Only

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: with 'Serious Game' to support the asthma treatment plan
  Interventions: Device: Serious Game (SG)
- Group 2: without 'Serious Game' and will follow the standard treatment plan

INTERVENTIONS:
Device: Serious Game (SG) — SG which was conceived as a running game, in which an Avatar runs through the forest and overcomes obstacles through the player's performance of physical exercises.
  Children will play while watching an imaginary Avatar, who shows the right movements to perform in order to collect rewards. SG will be projected with a 4K projector and controlled by the child's movements, which will be tracked in markerless mode using Azure's Kinect sensor. SG will include an adaptive tool to enable the experience based on the child's specific motor skills.
  The dynamics of SG will be adapted by considering real motor and physiological data acquired during each SG session via a wristband. These data are necessary to keep the child in the aerobic zone (60-80% of maximum heart rate). The movements are:
  1. Side bending: Moving an obstacle to open a passage.
  2. High jump: Overcoming a low, frontal obstacle.
  3. Side lunge: Avoiding a side obstacle.
  4. Squat: Passing under a low, frontal obstacle.
  Groups: Group 1

SUMMARY:
The main purpose of 'Serious Games' (SG) is to provide opportunities for constructive learning and training. They are well-accepted instruments in therapeutic interventions and have been found to be efficient to improve cognitive areas, social interaction and motor skill function.

The SG is expected to improve asthmatic children's behaviour by providing a positive psychosocial experience with positive effects on asthma outcomes.

Participants will be subjected to SG as part of routine medical care, and researchers will study the effect of SG.

The aim of the study is to evaluate the impact of an innovative SG on neurobehavioural patterns through a randomised controlled pilot study in adolescents with controlled asthma and on the modulation of the expression pattern of CTRA 'Conserved Transcriptional Response to Adversity'.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of controlled asthma according to GINA recommendations (http://ginasthma.org)

Exclusion Criteria:

* flare-ups requiring oral corticosteroids within the last four weeks
* use of leukotriene receptor antagonists or therapy as required in the last four weeks
* respiratory infections within the last four weeks
* immunological, metabolic, cardiac or neurological diseases
* obesity
* preterm birth
* major malformations of the respiratory system
* active smoking
* pregnancy

Ages: 12 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Male and female children aged 12 to 17 years. According to a computer-generated list, thirty children with controlled persistent asthma will be randomised into two groups: Asthma Group 1 and Asthma Group 2 'standard care'.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) | 6 months
  Questionnaires
Skills and Difficulties Questionnaire (SDQ-Ita) | 6 months

SECONDARY OUTCOMES:
Conserved Transcriptional Response to Adversity (CTRA) | 6 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uchida Y, Kitayama S, Akutsu S, Park J, Cole SW. Optimism and the conserved transcriptional response to adversity. Health Psychol. 2018 Nov;37(11):1077-1080. doi: 10.1037/hea0000675. Epub 2018 Sep 17. PMID 30221968
- [Background] Cole SW. The Conserved Transcriptional Response to Adversity. Curr Opin Behav Sci. 2019 Aug;28:31-37. doi: 10.1016/j.cobeha.2019.01.008. Epub 2019 Feb 25. PMID 31592179
- [Background] Mehl MR, Raison CL, Pace TWW, Arevalo JMG, Cole SW. Natural language indicators of differential gene regulation in the human immune system. Proc Natl Acad Sci U S A. 2017 Nov 21;114(47):12554-12559. doi: 10.1073/pnas.1707373114. Epub 2017 Nov 6. PMID 29109260
- [Background] Resztak JA, Farrell AK, Mair-Meijers H, Alazizi A, Wen X, Wildman DE, Zilioli S, Slatcher RB, Pique-Regi R, Luca F. Psychosocial experiences modulate asthma-associated genes through gene-environment interactions. Elife. 2021 Jun 18;10:e63852. doi: 10.7554/eLife.63852. PMID 34142656
- [Background] Ferrante G, Licari A, Marseglia GL, La Grutta S. Digital health interventions in children with asthma. Clin Exp Allergy. 2021 Feb;51(2):212-220. doi: 10.1111/cea.13793. Epub 2020 Dec 6. PMID 33238032
- [Background] Montalbano L, Ferrante G, Montella S, Cilluffo G, Di Marco A, Bozzetto S, Di Palmo E, Licari A, Leonardi L, Caldarelli V, Ghezzi M, La Grutta S, Rusconi F; Italian Pediatric Severe Asthma Network (IPSAN) Program of Italian Paediatric Respiratory Society (IPRS). Relationship between quality of life and behavioural disorders in children with persistent asthma: a Multiple Indicators Multiple Causes (MIMIC) model. Sci Rep. 2020 Apr 24;10(1):6957. doi: 10.1038/s41598-020-62264-9. PMID 32332757
- [Background] Montalbano L, Cilluffo G, Gentile M, Ferrante G, Malizia V, Cibella F, Viegi G, Passalacqua G, La Grutta S. Development of a nomogram to estimate the quality of life in asthmatic children using the Childhood Asthma Control Test. Pediatr Allergy Immunol. 2016 Aug;27(5):514-20. doi: 10.1111/pai.12571. Epub 2016 May 6. PMID 27018497
- [Background] Montella S, Baraldi E, Cazzato S, Aralla R, Berardi M, Brunetti LM, Cardinale F, Cutrera R, de Benedictis FM, di Palmo E, Di Pillo S, Fenu G, La Grutta S, Lombardi E, Piacentini G, Santamaria F, Ullmann N, Rusconi F; Italian Pediatric Severe Asthma Network (IPSAN) on behalf of the Italian Society of Pediatric Respiratory Diseases (SIMRI). Severe asthma features in children: a case-control online survey. Ital J Pediatr. 2016 Jan 22;42:9. doi: 10.1186/s13052-016-0217-z. PMID 26796331
- [Background] Ferrante G, La Grutta S. The Burden of Pediatric Asthma. Front Pediatr. 2018 Jun 22;6:186. doi: 10.3389/fped.2018.00186. eCollection 2018. PMID 29988370
- [Background] Waltz E. First video game to treat disease gains FDA okay. Nat Biotechnol. 2020 Nov;38(11):1224-1225. doi: 10.1038/s41587-020-0726-6. No abstract available. PMID 33144726
- [Background] Davis NO, Bower J, Kollins SH. Proof-of-concept study of an at-home, engaging, digital intervention for pediatric ADHD. PLoS One. 2018 Jan 11;13(1):e0189749. doi: 10.1371/journal.pone.0189749. eCollection 2018. PMID 29324745
- [Background] Licari A, Ferrante G, Marseglia Md GL, Corsello Md G, La Grutta S. What Is the Impact of Innovative Electronic Health Interventions in Improving Treatment Adherence in Asthma? The Pediatric Perspective. J Allergy Clin Immunol Pract. 2019 Nov-Dec;7(8):2574-2579. doi: 10.1016/j.jaip.2019.08.008. Epub 2019 Aug 16. PMID 31425835